CLINICAL TRIAL: NCT00076440
Title: Antigonadotropin-Leuprolide in Alzheimer's Disease Drug INvestigation (ALADDIN) VP 104 Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Voyager Pharmaceutical Corporation (Industry)
Organization: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IA0051
Record Dates: First submitted 2004-01-22; First posted 2004-01-26 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2007-03

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Leuprolide

INTERVENTIONS:
Drug: Leuprolide acetate

SUMMARY:
ALADDIN is a research study to investigate the safety and effectiveness of leuprolide (a hormone drug) to improve the cognitive function and slow the progression of Alzheimer's disease (AD) in men 65 years and older with mild to moderate Alzheimer's disease who reside in the community.

DETAILED DESCRIPTION:
ALADDIN is a clinical trial investigating the safety and effectiveness of leuprolide (a hormone drug) to improve the cognitive function and slow the progression of Alzheimer's disease (AD). The study will include treatment of men 65 years and older with mild to moderate Alzheimer's disease who reside in the community. The objective is to evaluate the safety and efficacy of two different doses of leuprolide to improve the cognitive function and slow the progression of AD, as measured by the ADAS-COG and the Clinical Global Impression (CGI). Measures of behavioral disturbances, and quality of life of the caregiver will be made also. The study design is randomized, double blind, placebo-controlled, parallel group design with a 2:1 randomization of drug to placebo. Sample size will include 90 participants from multiple test sites.

Following initial screening and baseline visits, the participant and caregiver will visit the site 8 times for a total of 10 visits over 48 weeks. The drug is administered via injection every 3 months. Safety assessments are completed and psychometric testing is done. Participant's memory, behavior, and global functioning are assessed during the participant and caregiver interviews. Each visit takes approximately 2 hours.

ELIGIBILITY:
Inclusion Criteria:

Patients who satisfy all of the inclusion criteria listed below will be eligible for entry into the trial.

* Patient and responsible caregiver can give their consent by signing the IRB-approved Informed Consent Form; or, when the patient is judged by the Investigator to be unable to give consent, the legally authorized representative gives consent by signing the consent form and the patient gives assent, in accord with local regulations;
* Male;
* 65 years of age or older;
* Diagnosis of probable AD according to the National Institute of Neurological Disorders-Alzheimer's Disease and Related Disorders Association (NINDS-ADRDA) criteria, and the Investigator ascertains that the condition was present at least 6 months prior to screening;
* Taking a drug for the treatment of AD, such as a cholinesterase inhibitor and/or Memantine®, which they began taking at least 90 days prior to baseline and, in the Investigator's opinion, the dosage will likely remain stable throughout the trial; or, they have never taken such a drug or stopped taking it at least 90 days prior to baseline and will likely refrain from taking such treatment throughout the trial;
* Taking other drugs or substances that have purported cognition-enhancing properties such as ginkgo biloba or Vitamin E, which they began taking at least 60 days prior to baseline and, in the Investigator's opinion, the dosage will likely remain stable throughout the trial; or, they have never taken such a drug or stopped taking it at least 90 days prior to baseline and will likely refrain from taking such treatment throughout the trial;
* Mini Mental State Examination (MMSE) score of 12 to 24 (inclusive) at the screening visit;
* Brain imaging study (CT scan, MRI or PET) performed at the time of their initial diagnosis of AD or after that time, and the findings were consistent with a diagnosis of probable AD, or, if a brain imaging study has not been performed, one will be performed during the screening process;
* Rosen Modified Hachinski score of 4 or lower at the screening visit, supporting the Investigator's clinical judgment that the patient's dementia is probable AD and not of vascular origin;
* Fluent in English or Spanish and completed at least 6 years of education;
* Live at home or in a congregate living facility for requirements other than skilled nursing care, and have a caregiver who sees the patient at least three times a week for a total of at least 10 hours and can sign the consent form, provide information pertinent to the patient's cognitive status, accompany the patient on clinic visits, and participate in the evaluations.
* Hamilton Depression Scale (17-item version) (HamD) score of 14 or less at the screening visit;
* DEXA scan, performed at screening, within normal limits (i.e., a T-score of greater than -2.0); or, if their DEXA measure was abnormally low (i.e., a T-score of -2.0 or lower), in either a lumbar vertebra or hip, to specifically include a T-score for the femoral neck), they were receiving treatment for osteoporosis/osteopenia for at least 3 weeks prior to baseline and that treatment is not expected to change during the course of the trial; or, if their DEXA measure was abnormally low and they are not receiving treatment for osteoporosis/osteopenia, they may proceed to baseline after 3 weeks of treatment for osteoporosis/osteopenia provided that all inclusion/exclusion criteria are met, including assessment of the HamD, concomitant medications, ECG and laboratory tests performed within 45 days of baseline show that they are eligible;
* Screening laboratory test values do not indicate significant medical conditions that would interfere with their participation in and completion of the study.

Exclusion criteria:

Patients with any of the exclusion criteria listed below will be ineligible for entry into the study.

* Female;
* Younger than 65 years of age;
* Significant neurological disease affecting the brain or psychiatric disease other than AD, such as major depression, schizophrenia, epilepsy, Parkinson's disease, or stroke;
* Current significant systemic illness or symptoms of organ failure;
* Screening ECG shows evidence of a serious and/or unstable condition or a recent (within 6 months) myocardial infarction as determined by the Investigator;
* PSA test result exceeds 4.0 ng/mL;
* Receiving testosterone;
* Taking a drug for the treatment of AD for less than 90 days prior to baseline; or, in the opinion of the Investigator, they are likely to either require a change in dose or discontinuation of the drug;
* Never received cholinesterase inhibitor treatment, and the likelihood of their starting such treatment during the study is other than low, or they have taken and discontinued cholinesterase inhibitor treatment in the past and the likelihood of their resuming cholinesterase inhibitor treatment during the study is other than low;
* Started or changed within 60 days prior to the screening visit the dosage of any drug (including OTC) that affects cognitive function, such as neuroleptics, antidepressants, anxiolytics, sedatives, hypnotics, anti-convulsants, centrally acting antihypertensive agents such as clonidine and Aldomet; or other medications that have been shown to have possible effects on cognition such as Vitamin E, nonsteroidal anti-inflammatory drugs, and statins, or if, in the Investigator's opinion, the dosage of such medication is likely to be changed during the course of this trial. Any changes in the dosage of any of these drugs during the course of the trial and the reason for the change must be fully recorded in the concomitant medication page of the patient's case report form (CRF). If a drug that affects cognition (e.g., a hypnotic or anxiolytic drug) is given on a PRN basis, such treatment should be interrupted for 12 hours before a visit, if possible;
* Taking coumadin or anti-Parkinsonian medications;
* Have taken other investigational drugs within 30 days or 5 half-lives prior to randomization, whichever is longer;
* Taking other medications known to affect serum gonadotropin (Gn) concentrations, such as goserelin or danazol;
* A screening HamD score of 15 or higher;
* Abuse or dependence on alcohol or other substances satisfies criteria for DSM-IV categories 303.9 or 305;
* Donated blood within 30 days of baseline or are likely to do so during the course of the trial;
* History of cancer, particularly breast cancer or known or suspected prostate cancer, within the last 5 years, except for basal cell or squamous cell cancer of the skin;
* Clinically significant bladder outlet obstruction, in the judgment of the Investigator or designated examining physician;
* Abnormalities of the esophagus which delay esophageal emptying such as stricture or achalasia, or are unable to stand or sit upright for at least 30 minutes;
* Sleep apnea.

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90
Dates: Start 2003-12; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard L. Bowen, MD, Principal Investigator — Voyager Pharmaceutical Corporation
Locations (13):
- United States (13):
  - Margolin Brain Institute, Fresno, California
  - Bay Area Research Institute, Lafayette, California
  - Southwest Clinical Research, Rancho Mirage, California
  - Geriatric and Adult Psychiatry LLC, Hamden, Connecticut
  - Baumel-Eisner Neuromedical Institute, Boca Raton, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Baumel-Eisner Neuromedical Institute, Fort Lauderdale, Florida
  - Baumel-Eisner Neuromedical Institute, Miami Beach, Florida
  - Meridien Research, St. Petersburg, Florida
  - Boston University School of Medicine, Boston, Massachusetts
  - Medical University of South Carolina, Charleston, South Carolina
  - Innovative Clinical Research Center, Alexandria, Virginia
  - Middleton VA Wisconsin Alzheimer's Institute, Madison, Wisconsin

REFERENCES:
- [Background] Bowen RL, Smith MA, Harris PL, Kubat Z, Martins RN, Castellani RJ, Perry G, Atwood CS. Elevated luteinizing hormone expression colocalizes with neurons vulnerable to Alzheimer's disease pathology. J Neurosci Res. 2002 Nov 1;70(3):514-8. doi: 10.1002/jnr.10452. PMID 12391612
- [Background] Short RA, Bowen RL, O'Brien PC, Graff-Radford NR. Elevated gonadotropin levels in patients with Alzheimer disease. Mayo Clin Proc. 2001 Sep;76(9):906-9. doi: 10.4065/76.9.906. PMID 11560301
- [Background] Bowen RL, Isley JP, Atkinson RL. An association of elevated serum gonadotropin concentrations and Alzheimer disease? J Neuroendocrinol. 2000 Apr;12(4):351-4. doi: 10.1046/j.1365-2826.2000.00461.x. PMID 10718932